CLINICAL TRIAL: NCT00151606
Title: Evaluation of Two Protocols to Prevent the Acquisition of Methicillin-Resistant Staphylococcus Aureus in Intensive Care Units.
Brief Title: Comparison of Two Protocols to Prevent the Acquisition of Methicillin-Resistant Staphylococcus Aureus.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Ministry of Health, France (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AFSSAPS 020551; PHRC/01-07; CIC0203/010
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2006-01-10 (Estimated); Status verified 2006-01

CONDITIONS: Nosocomial Infections; MRSA Colonization
Keywords: Infection prevention; Isolation; Resistant bacteria; MRSA colonization
MeSH Terms: conditions — Cross Infection

INTERVENTIONS:
Procedure: Reinforced isolation + Muciprocine

SUMMARY:
Nosocomial infections is a major problem in intensive care units due to both growing incidence and pathogens implicated which become increasingly resistant to antibiotics. According to the Center for Disease Control (USA), Staphylococcus aureus is responsible for approximately 10% of cases. In Europe, 79% of the S.aureus strains are resistant to methicillin, a routinely used antibiotic. Recommendations for the prevention of transmission of these resistant bacteria are rarely based on controlled trials. Therefore the aim of our study is to evaluate two protocols to prevent the acquisition of methicillin-resistant S. Aureus in intensive care units: either a reinforced isolation precautions protocol or a standard precautions protocol.

DETAILED DESCRIPTION:
Recommendations for the prevention of transmission of resistant bacteria in intensive care units (ICU) are rarely based on controlled trials. For this reason, we compared a reinforced isolation precautions protocol (RIPP) with a standard precautions protocol (SPP) for the acquisition of methicillin-resistant Staphylococcus aureus (MRSA) in 2 intensive care units.

Evaluation: the risk for MRSA carriage was defined on admission if 1 of 3 criteria were met: hospitalization in the past year, transfer with prior length of stay ≥2 days, prior history of MRSA in the 5 past years.

Intervention: Randomization 1/1 of a total of 500 patients to either protocol; MRSA screening was performed at the sites of carriage and colonization at inclusion, every week and at ICU discharge in all patients; the results were given to the clinicians only for the patients of the RIPP group.

Protocols: the SPP was consistent with the CDC recommendations and included transmission-based isolation precautions to patients with clinical samples involving resistant bacteria (including MRSA) or highly transmissible organisms. The RIPP included the extension of isolation precautions (1) to patients at risk for MRSA on admission until screening results proved negative and (2) to MRSA-positive patients on screening or clinical samples until further negative samples, in whom nasal mupirocin decontamination was added. Compliance with the recommendations of each protocol was controlled by an audit.

The efficacy is assessed on the proportion of patients who acquired MRSA at any site.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years
* Expected length of stay > 48h in intensive care unit
* Informed written consent

Exclusion Criteria:

* Cerebral death
* Care limitation
* Neutropenia
* Documented MRSA on admission
* Patients receiving antistaphylococcal topical antibiotics on admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2002-12; Study Completion 2004-02

PRIMARY OUTCOMES:
Proportion of patients who acquired MRSA at any site during their hospitalization in intensive care unit.

SECONDARY OUTCOMES:
- Rate of nosocomial MRSA infections
- Rate of nosocomial infections due to other pathogens
- Rate of nosocomial infections according to the site
- Death rate at the exit of intensive care unit
- Additional cost due to reinforced isolation protocol
- Antistaphylococcal antibiotics use in both protocols
- Number of days of antibiotherapy
- Time and cause of septic isolation

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Camus, MD, Principal Investigator — Rennes University Hospital; Eric Bellissant, MD, PhD, Study Chair — Rennes University Hospital
Locations (2):
- France (2):
  - Service de Maladies Infectieuses et Réanimation Médicale - Hôpital Pontchaillou, Rennes
  - Service de Réanimation Médicale - Hôpital Bretonneau, Tours

REFERENCES:
- [Background] Chaix C, Durand-Zaleski I, Alberti C, Brun-Buisson C. Control of endemic methicillin-resistant Staphylococcus aureus: a cost-benefit analysis in an intensive care unit. JAMA. 1999 Nov 10;282(18):1745-51. doi: 10.1001/jama.282.18.1745. PMID 10568647
- [Background] Girou E, Pujade G, Legrand P, Cizeau F, Brun-Buisson C. Selective screening of carriers for control of methicillin-resistant Staphylococcus aureus (MRSA) in high-risk hospital areas with a high level of endemic MRSA. Clin Infect Dis. 1998 Sep;27(3):543-50. doi: 10.1086/514695. PMID 9770155
- [Result] Camus C, Bellissant E, Sebille V, Perrotin D, Garo B, Legras A, Renault A, Le Corre P, Donnio PY, Gacouin A, Le Tulzo Y, Thomas R. Prevention of acquired infections in intubated patients with the combination of two decontamination regimens. Crit Care Med. 2005 Feb;33(2):307-14. doi: 10.1097/01.ccm.0000152224.01949.01. PMID 15699832
- [Derived] Camus C, Bellissant E, Legras A, Renault A, Gacouin A, Lavoue S, Branger B, Donnio PY, le Corre P, Le Tulzo Y, Perrotin D, Thomas R. Randomized comparison of 2 protocols to prevent acquisition of methicillin-resistant Staphylococcus aureus: results of a 2-center study involving 500 patients. Infect Control Hosp Epidemiol. 2011 Nov;32(11):1064-72. doi: 10.1086/662180. Epub 2011 Sep 29. PMID 22011532